CLINICAL TRIAL: NCT04262154
Title: SAABR: Single Arm Phase II Study of AR Targeted Therapy + Atezolizumab + GnRH Analog and Stereotactic Body Radiotherapy (SBRT) to the Prostate in Men With Newly Diagnosed Hormone-sensitive Metastatic Prostate Cancer
Brief Title: Study of Abiraterone Acetate or Enzalutamide, Atezolizumab, GnRH Analog and Radiation Therapy in Men With Newly Diagnosed Hormone-sensitive Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-461
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Prostate Cancer
Keywords: Abiraterone Acetate; Atezolizumab; GnRH Analog; Radiation Therapy; Hormone sensitive prostate cancer; Stereotactic Body Radiotherapy; SBRT; Metastatic prostate cancer; 19-461; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Prostatic Neoplasms | interventions — atezolizumab; abiraterone; Prednisone; Gonadotropin-Releasing Hormone; Radiosurgery; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metastatic Prostate Cancer (Experimental): Participants will have untreated metastatic (M1a/b/c) hormone-sensitive prostate cancer documented by positive bone scan or metastatic lesion on CT or MRI; untreated is defined as having never received surgical, radiotherapeutic, or systemic therapy for their prostate cancer.Group 1 and 2. The first 20 patients enrolled will be in Group 1 and the remaining patients (and those who are already on a GnRH analog) will be assigned to Group 2. All study participants will receive treatment with atezolizumab, abiraterone acetate, prednisone, GnRH analog, and SBRT, at the same doses.
  Interventions: Drug: Atezolizumab; Drug: Abiraterone; Drug: Prednisone; Drug: GnRH analog; Radiation: Stereotactic Body Radiotherapy (SBRT); Drug: Enzalutamide; Other: Follow up

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg IV over 60 minutes every 3 weeks
Drug: Abiraterone — Abiraterone 1000 mg daily
Drug: Prednisone — Prednisone 5 mg daily
Drug: GnRH analog — Any GnRH analog that is commercially available, injectable, and long acting analog of the native LHRH peptide and is administered to subjects via intramuscular injection. For this study, any GnRH analog can be used and thee manufacturer's instructions for dose and frequency should be followed.
Radiation: Stereotactic Body Radiotherapy (SBRT) — Intensity-modulated, image-guided, ultra-hypofractionated external beam radiotherapy (7.25-7.5 Gy x 5 to prostate and seminal vesicles QOD) will begin around 12 weeks (at Cycle 5 Day 1 (+/-5 days)
Drug: Enzalutamide — 160 mg once daily
Other: Follow up — Subjects who discontinue study treatment for reasons other than progression will be followed every 6 months (+/- 4 weeks) until a documented progression event (i.e., PSA, radiographic, or clinical progression). After a documented progressionevent (whether on treatment or during follow up), subjects will continue to be followed every 6 months (+/- 4 weeks) for overall survival via chart review and/or telephone call.

SUMMARY:
This study is to find out whether adding the study drug atezolizumab and stereotactic body radiotherapy (SBRT) to standard treatment with abiraterone acetate, prednisone, and Lupron® (leuprolide) is a safe and effective way to treat previously untreated metastatic prostate cancer, and to see whether the study treatment works better than the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide or have a legally authorized representative to provide written informed consent and HIPAA authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.

NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.

* Males 18 years of age and above
* Untreated metastatic (M1a/b/c) hormone-sensitive prostate cancer documented by positive bone scan or metastatic lesion on CT or MRI; untreated is defined as having never received surgical, radiotherapeutic, or systemic therapy to the prostate for cancer for their prostate cancer.

Note, 10 subjects who have had prior hormonal therapy (GnRH analog +/- first-generation anti-androgen such a bicalutamide) started up to 3 months prior to signing consent to the trial will be permitted to enroll onto the study if they have demonstrated a decline in PSA. Anti-androgens must be stopped prior to Cycle 1.

Note: patients who have started bicalutamide (Casodex) with or without a GnRH analog must stop prior to being registered on trial

* Biopsy-proven adenocarcinoma of the prostate
* Eligible for SBRT per institutional guidelines
* ECOG status of 0 or 1
* Normal organ function with acceptable initial laboratory values within 14 days of treatment start:

ANC ≥ 1,500 /µl Lymphocyte count ≥ 0.5 x 109/L (500/µL) Albumin ≥ 3.5 g/dL Hemoglobin ≥ 9 g/dL Platelet count ≥ 100,000 /µl Creatinine within institutional normal limits Potassium ≥ 3.5 mmol/L(within institutional normal range) Bilirubin ≤1.5 x ULN Patients with known Gilbert disease: serum bilirubin ≤3 x ULN)

SGOT(AST), SGPT ≥ 2.5 ULN with the following exceptions:

(ALT), and AST and (ALT), and Alkaline Phosphatase (ALP) Patients with documented liver metastases: AST and ALT ≤ 5 x ULN; Patients with documented liver or bone metastases: ALP ≤ 5 x ULN INR ≤ 1.5 x ULN

* Subjects must agree to use a medically acceptable method of birth control (e.g., spermicide in conjunction with a barrier such as a condom) or sexual abstinence for the duration of the study, including 150 days after the last dose of study drug. Sperm donation is prohibited during the study and for 30 days after the last dose of study drug. Female partners must use hormonal or barrier contraception unless postmenopausal or abstinent.

Exclusion Criteria:

* History of malignancy within 3 years prior to initiation of study treatment, except for malignancies with a negligible risk of metastasis of dead (e.g., 5-year OS rate >90%), such as non-melanoma skin carcinoma
* Pathological finding consistent with pure small cell carcinoma of the prostate
* Prostate volume > 80 cc
* Known or suspected brain metastasis or active leptomeningeal disease
* Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g. bone metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patient should be recovered from effects of radiation. There is no required minimum recovery period. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g.,epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment).
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (one monthly or more frequently).
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic BP ≥95 mmHg). Subjects with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Positive HIV test at screening
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test and/or HBV PCR at screening. Patients currently treated with anti-viral therapy for HBV. Subjects with a past or resolved HBV infection, defined as having a negative HBsAg and HBV PCR test and a positive total hepatitis B core antibody (HBcAb) test at screening, are eligible for the study.
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for subjects who have a positive HCV antibody test.
* History of adrenal dysfunction
* Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Subjects with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone
  * Subjects with controlled Type 1 diabetes mellitus who are on an insulin regimen
  * Subjects with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., subjects with psoriatic arthritis are excluded) are allowed provided all the following conditions are met:
* Rash must cover < 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, cerebrovascular accident, unstable arrhythmia or unstable angina) within 6 months prior to initiation of study treatment
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Prior allogeneic stem cell or solid organ transplantation

  * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-a agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Subjects who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Sponsor Principal Investigator approval has been obtained.
  * Subjects who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the abiraterone or prednisone formulations
* Any other disease, metabolic dysfunction, physical examination finding, clinical laboratory finding or situation that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Failure-free rate at 2 years | 2 years
  Failure is defined as: biochemical failure, radiographic progression defined by PCWG3, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org